CLINICAL TRIAL: NCT01180985
Title: Dispensing Evaluation of a Galyfilcon A Prototype Lens and a Marketed Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-1636BD
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- galyfilcon A prototype/comfilcon A (Other): The galyfilcon A prototype lenses are worn during first period and comfilcon A lenses worn during second period. Each period consists of daily lens wear for one week.
  Interventions: Device: galyfilcon A prototype lens; Device: comfilcon A
- comfilcon A/galyfilcon A prototype (Other): The comfilcon A lenses are worn during first period and galyfilcon A prototype lenses worn during second period. Each period consists of daily lens wear for one week.
  Interventions: Device: galyfilcon A prototype lens; Device: comfilcon A

INTERVENTIONS:
Device: galyfilcon A prototype lens — silicone hydrogel contact lens
Device: comfilcon A — silicone hydrogel contact lens
  Other Names: Biofinity® contact lens

SUMMARY:
The purpose of this study is to compare visual acuity and redness of eyes between a prototype contact lens and an already marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a current spherical soft contact lens wearer and willing to wear the study lenses on a daily wear basis for the duration of the study.
* The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 5.00D.
* Any cylinder power must be ≤ -0.75D.
* The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2010-07-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Jacksonville, Florida
  - Orlando, Florida
  - Fincastle, Virginia
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a four (4) site, bilateral crossover study. Data were collected in three (3) visits (initial, 1 wk follow-up, and final visit).
Pre-assignment Details: Fifty-three (53) subjects enrolled, one(1) subject was discontinued and fifty-two (52) completed the study.
Groups:
- Galyfilcon A (Test)/Comfilcon A (Control); Comfilcon A (Control)/Galyfilcon A (Test): Each subject wore the assigned lens type for 7 +/- 1 days, according to the randomization scheme.
Period: Period 1 (7 +/- Days)
Arm/Group | Galyfilcon A (Test)/Comfilcon A (Control) | Comfilcon A (Control)/Galyfilcon A (Test)
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0
Period: Period 2 (7 +/- 1 Days)
Arm/Group | Galyfilcon A (Test)/Comfilcon A (Control) | Comfilcon A (Control)/Galyfilcon A (Test)
Started | 27 | 26
Completed | 26 | 26
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All enrolled subjects at baseline.
Arm/Group | All Subjects
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.00 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Monocular
Description: Snellen monocular visual acuity measurement was measured in both eyes that wore lenses for one week and came in for the evaluation with an inserted lens.
Time Frame: after 7 +/- 1 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Comfilcon A Lens (Control): All eyes of subjects who wore comfilcon A lenses for 7 +/-1 days to the time of evaluation
- Galyfilcon A Lens (Test): All eyes of subjects who wore galyfilcon A lenses for 7 +/- 1 days to the time of evaluation
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 52 | 52
Number analyzed (eyes) | 104 | 104
eyes
  20/15 monocular | 53 | 49
  20/20 monocular | 49 | 48
  20/25 monocular | 2 | 4
  20/30 monocular | 0 | 3

2. Primary Outcome: Visual Acuity Binocular
Description: Snellen binocular visual acuity measurement
Time Frame: after 7 +/- 1 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: participants
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 52 | 52
participants
  20/10 binocular | 0 | 1
  20/15 binocular | 31 | 29
  20/20 binocular | 21 | 20
  20/25 binocular | 0 | 1
  20/30 binocular | 0 | 1

3. Primary Outcome: Subjective Assessment of Lens Comfort Using the Contact Lens User Experience (CLUE)TM Questionnaire.
Description: The contract Lens Experience (CLUE)TM questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: after 7 +/-1 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE score
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 50 | 50
CLUE score | 57.72 (4.47) | 67.06 (4.50)

4. Secondary Outcome: Limbal Redness
Description: Scale of 0 to 4, where 0=None, 2=Trace, 3=Mild, 4=Moderate, 5=Severe.
Time Frame: after 7 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 52 | 52
Number analyzed (eyes) | 104 | 104
eyes
  Grade 0 = No redness | 37 | 36
  Grade 1 = Trace redness | 36 | 42
  Grade 2 = Mild redness | 31 | 26

5. Primary Outcome: Subjective Assessment of Quality of Vision Using the Contact Lens User Experience(CLUE)TM Questionnaire.
Description: Contact Lens User Experience CLUE)TM questionnaire: A validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: after 7 +/- 1 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE score
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 50 | 50
CLUE score | 62.75 (2.83) | 59.98 (2.81)

6. Secondary Outcome: Bulbar Redness
Description: Scale of 0 to 4, where 0=None, 2=Trace, 3=Mild, 4=Moderate, 5=Severe.
Time Frame: after 7 days of lens wear
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 52 | 52
Number analyzed (eyes) | 104 | 104
eyes
  Grade 0 = No redness | 39 | 37
  Grade 1 = Trace redness | 55 | 59
  Grade 2 = Mild redness | 10 | 8

7. Secondary Outcome: Subjective Assessment of Lens Comfort Using the Contact Lens User Experience (CLUE)TM Questionnaire.
Description: as for outcome 5
Time Frame: 10 minutes after lens insertion at time of initial lens fitting
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: CLUE score
Groups:
- Comfilcon A Lens (Control): All subjects who wore comfilcon A lenses
- Galyfilcon A Lens (Test): All subjects who wore galyfilcon A lenses
Arm/Group | Comfilcon A Lens (Control) | Galyfilcon A Lens (Test)
Number analyzed (Participants) | 50 | 50
CLUE score | 80.32 (18.36) | 82.76 (17.01)

ADVERSE EVENTS:
Groups:
- Galyfilcon A Prototype/Comfilcon A: All enrolled subjects were to wear both lenses through the course of the study.
Arm/Group | Galyfilcon A Prototype/Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written consent from the Sponsor.